CLINICAL TRIAL: NCT04205890
Title: Intravenous Ketamine Effects on Functional Neuroanatomy
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor is no longer interested in funding the study
Sponsor: Neurological Associates of West Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20190792
Record Dates: First submitted 2019-12-16; First posted 2019-12-20 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Depression
Keywords: intravenous ketamine; treatment-resistant depression
MeSH Terms: conditions — Depression; Depressive Disorder, Treatment-Resistant | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: The purpose of this study is to investigate the neuroanatomical effects of ketamine treatment on patients with treatment-resistant depression. We will compare the neuroimaging of patients several days before and after injection in order to assess the more durable changes induced by ketamine. We will analyze changes in perfusion, neurovascular coupling, and functional connectivity that are correlated with psychiatric measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ketamine (Experimental): The present study is designed as a prospective data analysis of patient response to the use of ketamine to treat treatment-resistant depression. For Phase I trail, 10 patients of any gender with an age range of 18 to 70 who have undergone the outlined procedure will be recruited for inclusion. A week before the scheduled ketamine treatment, the patients will have fMRI scans, including structural T1, Arterial Spin Labeling, and Resting BOLD. The scans take around 30 minutes at no charge to the patients. The ketamine will be injected per the doctor's orders to achieve a dissociative state; dosage will vary (see below) depending on every individual's unique treatment plan. The same scans will be taken two days after treatment.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — The ketamine will be injected per the doctor's orders to achieve a dissociative state; dosage varies between 75mg - 1000mg depending on every individual's unique treatment plan.

SUMMARY:
The purpose of this study is to investigate the neuroanatomical effects of ketamine treatment on patients with treatment-resistant depression. The investigators will compare the neuroimaging of patients several days before and after injection in order to assess the more durable changes induced by ketamine. In addition, changes in perfusion will be analyzed, in addition to changes in neurovascular coupling, and functional connectivity that are correlated with psychiatric measures.

DETAILED DESCRIPTION:
The present study is designed as a prospective data analysis of patient response to the use of ketamine to treat treatment-resistant depression. For Phase I trail, 10 patients of any gender with an age range of 18 to 70 who have undergone the outlined procedure will be recruited for inclusion. Patients will be examined by the principle investigator. All patients must be diagnosed with persistent treatment-resistant depression and prescribed ketamine. Patients will be accepted regardless of if the depression coincided with anxiety and/or pain. Patient status will be assessed using the Beck Depression Inventory, Beck Anxiety Inventory, and Brief Pain Inventory. Patients must have a Beck Depression Inventory score of 10 or above. These scores will be used as baseline data. Patients will be offered the option of participating in the study and provided informed consent for neuroimaging before and after the ketamine treatment.

A week before the scheduled ketamine treatment, the patients will have fMRI scans, including structural T1, Arterial Spin Labeling, and Resting BOLD. The scans take around 30 minutes at no charge to the patients. The ketamine will be injected per the doctor's orders to achieve a dissociative state; dosages varies between 75mg - 1000mg depending on every individual's unique treatment plan. The same scans will be taken two days after treatment.

ELIGIBILITY:
Inclusion Criteria:

* In order for a subject to be considered for this study, the patient must have been diagnosed with treatment-resistant depression, meaning the patient failed three medications and has been suffering from moderate treatment-resistant depression for over 6 months, indicated by a Beck Depression Inventory score of 10 or above. The patient must have been prescribed ketamine as part of their treatment plan, completely independent of any research. The patient must be willing to comply with the study protocol.

Exclusion Criteria:

* In order for a subject to be considered for this study, he/she may not have any of the following:

  * Advanced stages of any terminal illness or any active cancer that requires chemotherapy
  * Hepatic impairment
  * Significant cytopenia
  * Cardiovascular, cerebrovascular, and peripheral vascular arterial thrombosis
  * Women who are pregnant, may become pregnant, or are breastfeeding
  * Any counter indications to ketamine
  * Subjects unable to give informed consent or in vulnerable categories, such as prisoners

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-02 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-05-28 (Actual)

PRIMARY OUTCOMES:
fMRI T1 baseline | Images to be acquired 7 days prior to Ketamine intervention
  T1-data was collected as a sagittal MPRAGE sequence. T1 images are corrected for field biasing and then skull stripped and linearly registered to standard MNI space. Each patients' T1 image is segmented into 100 cortical and 15 subcortical areas using the Harvard-Oxford Cortical and Subcortical structural atlas. Mean volume is computed for each of these regions for each patient, which can be used for quantitative comparison.
fMRI T1 post-intervention comparison | Images to be acquired at 2 days post-treatment
  T1-data was collected as a sagittal MPRAGE sequence. T1 images are corrected for field biasing and then skull stripped and linearly registered to standard MNI space. Each patients' T1 image is segmented into 100 cortical and 15 subcortical areas using the Harvard-Oxford Cortical and Subcortical structural atlas. Mean volume is computed for each of these regions for each patient, which can be used for quantitative comparison.
Arterial Spin Labeling (fMRI) baseline | Images to be acquired 7 days prior to Ketamine intervention
  Pulsed Arterial Spin Labeling is collected as an echo planar sequence. ASL data is superimposed over the acquired T1-weighted brain image demonstrating a map of cerebral perfusion. Quantification to CBF values (milliliters of blood per 100g of tissue per minute) is implemented and voxel-based comparisons showing perfusion values relative to the acquired data range are used for quantification.
Arterial Spin Labeling (fMRI) post-intervention comparison | Images to be acquired at 2 days post-treatment
  Pulsed Arterial Spin Labeling is collected as an echo planar sequence. ASL data is superimposed over the acquired T1-weighted brain image demonstrating a map of cerebral perfusion. Quantification to CBF values (milliliters of blood per 100g of tissue per minute) is implemented and voxel-based comparisons showing perfusion values relative to the acquired data range are used for quantification.
fMRI Resting Bold baseline | Images to be acquired 7 days prior to Ketamine intervention
  The signal change measured in BOLD imaging comes from the brain oversupplying the region of activation with oxygen, leading to a focal decrease in deoxygenated hemoglobin. Processed BOLD imaging allows for visualization of hemodynamic response (HR) and neurovascular coupling (NVC) based on signal variability and distribution. These elements can be quantified and used for comparison.
fMRI Resting Bold post-intervention comparison | Images to be acquired at 2 days post-treatment
  The signal change measured in BOLD imaging comes from the brain oversupplying the region of activation with oxygen, leading to a focal decrease in deoxygenated hemoglobin. Processed BOLD imaging allows for visualization of hemodynamic response (HR) and neurovascular coupling (NVC) based on signal variability and distribution. These elements can be quantified and used for comparison.

SECONDARY OUTCOMES:
Beck Depression Inventory | 7 days prior to treatment
  The BDI-II is a 21-question multiple-choice self-report inventory. Each question involves four possible responses, ranging in intensity from "0" (this item does not apply) to "3" (this item applies severely). The test is scored as the sum of all of the response values; this number is used to determine the severity of depressive symptoms. A score of 0 to 3 is possible for each question with a maximum total score of 63 points. The standard cutoff scores are as follows: 0-13 total points = minimal depression; 14-19 total points = mild depression; 20-28 total points = moderate depression; and 29-63 total points = severe depression. A reduction in the total score by at least 30% is considered to be clinically significant.
Beck Depression Inventory | Day of treatment
  The BDI-II is a 21-question multiple-choice self-report inventory. Each question involves four possible responses, ranging in intensity from "0" (this item does not apply) to "3" (this item applies severely). The test is scored as the sum of all of the response values; this number is used to determine the severity of depressive symptoms. A score of 0 to 3 is possible for each question with a maximum total score of 63 points. The standard cutoff scores are as follows: 0-13 total points = minimal depression; 14-19 total points = mild depression; 20-28 total points = moderate depression; and 29-63 total points = severe depression. A reduction in the total score by at least 30% is considered to be clinically significant.
Beck Depression Inventory | 2 days after treatment
  The BDI-II is a 21-question multiple-choice self-report inventory. Each question involves four possible responses, ranging in intensity from "0" (this item does not apply) to "3" (this item applies severely). The test is scored as the sum of all of the response values; this number is used to determine the severity of depressive symptoms. A score of 0 to 3 is possible for each question with a maximum total score of 63 points. The standard cutoff scores are as follows: 0-13 total points = minimal depression; 14-19 total points = mild depression; 20-28 total points = moderate depression; and 29-63 total points = severe depression. A reduction in the total score by at least 30% is considered to be clinically significant.
Beck Anxiety Inventory | 7 days prior to treatment
  The BAI is a 21-question multiple-choice self-report inventory that is used for measuring the severity of anxiety symptoms. Each of the 21 items asks whether the patient has experienced various anxiety symptoms in the last two weeks, and if so, how severely. Each question/answer is scored on a scale value of "0" (not at all) to "3" (severely). Higher total scores indicate more severe anxiety symptoms. The maximum total score possible is 63 points. The standard cutoff scores are: 0-7 = minimal anxiety; 8-15 = mild anxiety; 16-25 = moderate anxiety; 26-63 = severe anxiety. A reduction in score by at least 30% is considered clinically meaningful.
Beck Anxiety Inventory | Day of treatment
  The BAI is a 21-question multiple-choice self-report inventory that is used for measuring the severity of anxiety symptoms. Each of the 21 items asks whether the patient has experienced various anxiety symptoms in the last two weeks, and if so, how severely. Each question/answer is scored on a scale value of "0" (not at all) to "3" (severely). Higher total scores indicate more severe anxiety symptoms. The maximum total score possible is 63 points. The standard cutoff scores are: 0-7 = minimal anxiety; 8-15 = mild anxiety; 16-25 = moderate anxiety; 26-63 = severe anxiety. A reduction in score by at least 30% is considered clinically meaningful.
Beck Anxiety Inventory | 2 days after treatment
  The BAI is a 21-question multiple-choice self-report inventory that is used for measuring the severity of anxiety symptoms. Each of the 21 items asks whether the patient has experienced various anxiety symptoms in the last two weeks, and if so, how severely. Each question/answer is scored on a scale value of "0" (not at all) to "3" (severely). Higher total scores indicate more severe anxiety symptoms. The maximum total score possible is 63 points. The standard cutoff scores are: 0-7 = minimal anxiety; 8-15 = mild anxiety; 16-25 = moderate anxiety; 26-63 = severe anxiety. A reduction in score by at least 30% is considered clinically meaningful.
Brief Pain Inventory | 7 days prior to treatment
  Self-report measure containing a composite pain score and functional interference score. The pain subscale contains 4 questions, each with answers ranging from 0 'no pain' to 10 'pain as bad as you can imagine.' Total possible score for the pain subscale is 40 points. The functional/interference subscale contains 7 questions, with each answer ranging from 0 'does not interfere' to 10 'completely interferes.' The maximum possible score for the interference subscale is 70 points. The total overall composite BPI score is out of 100 maximum points. A clinical improvement is considered a decrease in BPI overall composite score by at least 30% from baseline.
Brief Pain Inventory | Day of Treatment
  Self-report measure containing a composite pain score and functional interference score. The pain subscale contains 4 questions, each with answers ranging from 0 'no pain' to 10 'pain as bad as you can imagine.' Total possible score for the pain subscale is 40 points. The functional/interference subscale contains 7 questions, with each answer ranging from 0 'does not interfere' to 10 'completely interferes.' The maximum possible score for the interference subscale is 70 points. The total overall composite BPI score is out of 100 maximum points. A clinical improvement is considered a decrease in BPI overall composite score by at least 30% from baseline.
Brief Pain Inventory | 2 days post-treatment
  Self-report measure containing a composite pain score and functional interference score. The pain subscale contains 4 questions, each with answers ranging from 0 'no pain' to 10 'pain as bad as you can imagine.' Total possible score for the pain subscale is 40 points. The functional/interference subscale contains 7 questions, with each answer ranging from 0 'does not interfere' to 10 'completely interferes.' The maximum possible score for the interference subscale is 70 points. The total overall composite BPI score is out of 100 maximum points. A clinical improvement is considered a decrease in BPI overall composite score by at least 30% from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Jordan, MD, Principal Investigator — The Neurological Associates of West Los Angeles; Taylor Kuhn, PhD, Principal Investigator — The Neurological Associates of West Los Angeles
Locations (1):
- Neurological Associates of West Los Angeles, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No
Data from this study will not be made publicly available due to ethical and privacy concerns. Anonymized data will be available upon reasonable request from any qualified investigator.

REFERENCES:
- [Background] Berman RM, Cappiello A, Anand A, Oren DA, Heninger GR, Charney DS, Krystal JH. Antidepressant effects of ketamine in depressed patients. Biol Psychiatry. 2000 Feb 15;47(4):351-4. doi: 10.1016/s0006-3223(99)00230-9. PMID 10686270
- [Background] Deakin JF, Lees J, McKie S, Hallak JE, Williams SR, Dursun SM. Glutamate and the neural basis of the subjective effects of ketamine: a pharmaco-magnetic resonance imaging study. Arch Gen Psychiatry. 2008 Feb;65(2):154-64. doi: 10.1001/archgenpsychiatry.2007.37. PMID 18250253
- [Background] Fava M. Diagnosis and definition of treatment-resistant depression. Biol Psychiatry. 2003 Apr 15;53(8):649-59. doi: 10.1016/s0006-3223(03)00231-2. PMID 12706951
- [Background] Lepine JP, Briley M. The increasing burden of depression. Neuropsychiatr Dis Treat. 2011;7(Suppl 1):3-7. doi: 10.2147/NDT.S19617. Epub 2011 May 31. PMID 21750622
- [Background] Maeng S, Zarate CA Jr, Du J, Schloesser RJ, McCammon J, Chen G, Manji HK. Cellular mechanisms underlying the antidepressant effects of ketamine: role of alpha-amino-3-hydroxy-5-methylisoxazole-4-propionic acid receptors. Biol Psychiatry. 2008 Feb 15;63(4):349-52. doi: 10.1016/j.biopsych.2007.05.028. Epub 2007 Jul 23. PMID 17643398
- [Background] Mayberg HS, Lozano AM, Voon V, McNeely HE, Seminowicz D, Hamani C, Schwalb JM, Kennedy SH. Deep brain stimulation for treatment-resistant depression. Neuron. 2005 Mar 3;45(5):651-60. doi: 10.1016/j.neuron.2005.02.014. PMID 15748841
- [Background] U.S. Department of Health and Human Services, National Institutes of Health, National Institute of Mental Health. (2019). Major Depression. Retrieved from https://www.nimh.nih.gov/health/statistics/major-depression.shtml
- [Background] U.S. Department of Health and Human Services, National Institutes of Health, National Institute of Mental Health. (2018). Depression. Retrieved from https://www.nimh.nih.gov/health/topics/depression/index.shtml